CLINICAL TRIAL: NCT05673681
Title: Registro de Melanoma de la AEDV
Brief Title: Spanish Academy of Dermatology and Venereology (AEDV) Melanoma Registry
Status: Recruiting | Type: Observational
Sponsor: Fundación Academia Española de Dermatología (Other)
Responsible Party: Sponsor
Other Study IDs: FAE-MEL-2022-01
Record Dates: First submitted 2023-01-02; First posted 2023-01-06 (Actual); Last update posted 2023-01-09 (Actual); Status verified 2023-01

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this patient registry is to describe risk factors for bad prognosis of melanoma in Spain. The main questions it aims to answer are:

* To describe socioeconomical individual risk factors associated with melanoma prognosis, such as gender, residence area or socioeconomic level.
* To describe potentially modifiable characteristics of health care associated with prognosis, such as waiting times, type of centre that makes the diagnosis or use of teledermatology Participants data will be gathered for analysis, without any change in the way that they are being treated.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive patients with a diagnosis of invasive primary cutaneous melanoma in participating centres.

Exclusion Criteria:

* In-situ melanomas
* non-cutaneous melanomas,
* metastatic melanoma with unknown primary site.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All consecutive patients with a diagnosis of invasive primary cutaneous melanoma in participating centres.
Sampling Method: Non-Probability Sample
Enrollment: 7000 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2032-06-01 (Estimated); Study Completion 2032-06-01 (Estimated)

PRIMARY OUTCOMES:
AJCC (American Joint Committee on Cancer) TNM stage (Tumor, node, metastasis) | 1 day At diagnosis
  Staging based on tumor thickness and ulceration, spread to lymph nodes and spread to distant sites.
Breslow thickness | 1 day At diagnosis
  Breslow thickness is the measurement of the depth of the melanoma from the surface of your skin down through to the deepest point of the tumour.

SECONDARY OUTCOMES:
Time to progression | through study completion, an average of 3 years
Survival | through study completion, an average of 3 years

CONTACTS AND LOCATIONS:
Locations (21):
- Spain (21):
  - Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona
  - Complexo Hospitalario Universitario de A Coruña, A Coruña
  - Hospital Clinic, Barcelona
  - Hospital San Juan de Dios, Córdoba
  - Hospital Universitario de Gran Canaria Dr Negrín, Las Palmas
  - Complejo Asistencial Universitario de León, León
  - Clínica Dermatológica Internacional, Madrid
  - Clínica Universitaria de Navarra ( sede de Madrid), Madrid
  - Hospital Clínico San Carlos, Madrid
  - Hospital La Paz, Madrid
  - Hospital Puerta de Hierro Majadahonda, Madrid
  - Ruber Internacional, Madrid
  - Hospital Central de Asturias, Oviedo
  - Hospital Son LLàtzer, Palma de Mallorca
  - Complexo Hospitalario Universitario de Pontevedra, Pontevedra
  - H.U. Nuestra Señora de la Candelaria, Santa Cruz de Tenerife
  - Hospital Universitario Virgen Macarena de Sevilla, Seville
  - Quirón Salud Sevilla, Seville
  - Hospital La Fé, Valencia
  - Instituto Valenciano de Oncología, Valencia
  - Hospital Miguel Servet, Zaragoza

IPD SHARING:
Plan to Share IPD: No